CLINICAL TRIAL: NCT03068611
Title: Development and Pilot Testing of a Multimodal Web-based Program to Address Heavy Drinking During Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Truth Initiative (Other)
Responsible Party: Principal Investigator, Christopher W. Kahler, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34AA024593 (NIH)
Record Dates: First submitted 2017-02-23; First posted 2017-03-03 (Actual); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Smoking Cessation; Alcohol Drinking
MeSH Terms: conditions — Smoking Cessation; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Web-based Smoking Cessation (Active Comparator): A website and text messaging program that is publicly available through BecomeAnEX.com. Participants have access to the website whenever they wish.
  Interventions: Behavioral: Standard Web-based Smoking Cessation
- Alcohol-focused Web-Based Smoking Cessation (Experimental): A modified version of the website and text messaging program that is publicly available through BecomeAnEX.com. This version includes specific information and feedback on alcohol use, allows participants to consider benefits of changing drinking, plans for changing drinking, and strategies. Participants have access to the website whenever they wish.
  Interventions: Behavioral: Alcohol-focused Web-Based Smoking Cessation

INTERVENTIONS:
Behavioral: Standard Web-based Smoking Cessation — A website and text messaging program that is publicly available through BecomeAnEX.com. Participants have access to the website whenever they wish.
  Arms: Standard Web-based Smoking Cessation
Behavioral: Alcohol-focused Web-Based Smoking Cessation — A website and text messaging program that is publicly available through BecomeAnEX.com. Participants have access to the website whenever they wish.
  Arms: Alcohol-focused Web-Based Smoking Cessation

SUMMARY:
The overall objective of this project is to develop and pilot-test a web-based smoking cessation program that specifically addresses heavy drinking (HD). The project builds upon a well-established, free evidence-based smoking cessation website, BecomeAnEX.org ("EX"), which is supported by Truth Initiative, a national non-profit public health organization, and its research arm, the Schroeder Institute. Investigators will develop an alternative version of BecomenAnEX that will include detailed content on alcohol's relation to smoking relapse, health effects of alcohol (including moderate drinking recommendations) along with related worksheets, feedback materials, and links to resources for drinking. Once a version of BecomeAnEX is developed that specifically addresses HD (called EX-HD), the investigators will conduct a one-arm open pilot of the site with 30 HD smokers recruited from newly registered BecomeAnEX users. The study will gather participant feedback on the site as well as site use metrics (e.g., number of logins, number of pages viewed, use of interactive components) and will revise EX-HD in response to this feedback in preparation for Stage 1b work. Stage 1b will use the updated EX-HD version to run a small scale randomized clinical trial where 120 participants will be randomly assigned to the standard version of BecomeAnEX or to EX-HD.

ELIGIBILITY:
Inclusion Criteria:

1. current daily smoking of at least one cigarette per day
2. meeting NIAAA criteria for past month heavy or at-risk drinking (for women: drinking 8+ drinks per week or consuming 4+ drinks on one occasion at least once in the past month; for men: drinking 15+ drinks per week or consuming 5+ drinks on one occasion at least once in the past month)
3. age 18 or older
4. willingness to provide contact and mailing information following consent

Exclusion Criteria:

1. history of severe alcohol withdrawal as indicated by past alcohol-induced seizures or delirium tremens;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Alcohol and Addiction Studies, Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kahler CW, Cohn AM, Costantino C, Toll BA, Spillane NS, Graham AL. A Digital Smoking Cessation Program for Heavy Drinkers: Pilot Randomized Controlled Trial. JMIR Form Res. 2020 Jun 8;4(6):e7570. doi: 10.2196/formative.7570. PMID 32348286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment was conducted online over 7 weeks (May to July, 2017). Only newly registered users of BecomeAnEX.org were recruited.
Period: Overall Study
Arm/Group | Standard Web-based Smoking Cessation | Alcohol-focused Web-Based Smoking Cessation
Started | 61 | 58
Completed | 30 (This is the number of participants followed through 6 months from enrollment.) | 33 (This is the number of participants followed through 6 months from enrollment.)
Not Completed | 31 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Web-based Smoking Cessation | Alcohol-focused Web-Based Smoking Cessation | Total
Number analyzed (Participants) | 61 | 58 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (12.9) | 37.1 (10.6) | 38.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 83
  Male | 19 | 17 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 60 | 55 | 115
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 50 | 48 | 98
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported 7-day Point-prevalence Smoking Abstinence at 1 Month
Description: Self-report abstinence from smoking
Time Frame: 1 month after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Web-based Smoking Cessation | Alcohol-focused Web-Based Smoking Cessation
Number analyzed (Participants) | 61 | 58
Participants | 10 | 10
Statistical Analysis 1: Comparison: Standard Web-based Smoking Cessation vs Alcohol-focused Web-Based Smoking Cessation; Test type: Superiority; p = .90, Chi-squared

2. Primary Outcome: Number of Participants Who Reported 7-day Point-prevalence Smoking Abstinence at 6 Months
Description: Self-report abstinence from smoking
Time Frame: 6 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Web-based Smoking Cessation | Alcohol-focused Web-Based Smoking Cessation
Number analyzed (Participants) | 61 | 58
Participants | 9 | 11
Statistical Analysis 1: Comparison: Standard Web-based Smoking Cessation vs Alcohol-focused Web-Based Smoking Cessation; Test type: Superiority; p = .54, Chi-squared

3. Primary Outcome: Number of Heavy Drinking Days at 1 Month
Description: Self reported number of days (in the past 30 days) drinking 4+/5+ drinks for women/men
Time Frame: 1 month after enrollment
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard Web-based Smoking Cessation | Alcohol-focused Web-Based Smoking Cessation
Number analyzed (Participants) | 45 | 40
Days | 2.9 (4.7) | 4.4 (6.3)
Statistical Analysis 1: Comparison: Standard Web-based Smoking Cessation vs Alcohol-focused Web-Based Smoking Cessation; Test type: Superiority; p = .36, t-test, 2 sided; Data were log-transformed transformed due to positive skewness

4. Primary Outcome: Number of Heavy Drinking Days at 6 Months
Description: Self reported number of days (in the past 30 days) drinking 4+/5+ drinks for women/men
Time Frame: 6 months after enrollment
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard Web-based Smoking Cessation | Alcohol-focused Web-Based Smoking Cessation
Number analyzed (Participants) | 30 | 33
Days | 2.6 (3.5) | 3.8 (6.7)
Statistical Analysis 1: Comparison: Standard Web-based Smoking Cessation vs Alcohol-focused Web-Based Smoking Cessation; Test type: Superiority; p = .92, t-test, 2 sided; Data were log-transformed to correct positive skewness

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Standard Web-based Smoking Cessation | Alcohol-focused Web-Based Smoking Cessation
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/58
Other Adverse Events (participants affected / at risk) | 0/61 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03068611/SAP_000.pdf
  • Study Protocol (2016-01-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT03068611/Prot_001.pdf